CLINICAL TRIAL: NCT03128541
Title: Influence of Body Positioning on the Identification of Tuffier's Line Using the Traditional Palpation Method: An Ultrasound Study.
Brief Title: Influence of Body Positioning on the Identification of Tuffier's Line Using the Palpation Method: An Ultrasound Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 218764
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ultrasound Spine in sitting position: Participants will be assigned to a sitting decubitus position to identify the Tuffier's Line
  Interventions: Diagnostic Test: Ultrasound spine
- Ultrasound Spine in lateral position: Participants will be assigned to a lateral decubitus position to identify the Tuffier's Line
  Interventions: Diagnostic Test: Ultrasound spine

INTERVENTIONS:
Diagnostic Test: Ultrasound spine — A ultrasound of the lumbar spine of each patient will be performed in both positions to identify vertebral levels

SUMMARY:
The study aims to ascertain whether being placed in a sitting or lateral decubitus position, influences identification of the midpoint of the L4/L5 intervertebral space, using manual demarcation of Tuffier's line. Participants will be randomly assigned to a sitting or lateral decubitus position. The mid-point of the L4/L5 intervertebral space will be identified using anatomical palpation and compared to the "true" mid-point measured by ultrasound. The procedure will be repeated in both positions on the same participant.The study will be a prospective, randomized, double blinded, crossover trial

DETAILED DESCRIPTION:
Anaesthetists insert epidurals or spinal anaesthetics (collectively called central neuraxial blocks) to patients during childbirth to provide pain relief and anaesthesia. A spinal anaesthetic involves the injection of pain relieving medicines directly into the sac of fluid that surrounds the spinal cord. An epidural uses a different technique to place a thin plastic tube into the fatty tissues that surround this sac. Spinal anaesthesia must be placed below where the spinal cord ends to avoid nerve trauma. Doctors have traditionally been taught to identify a safe level, by feeling the top of a patients hips and drawing an imaginary line between these two points across the patients back known as Tuffier's line. This identifies L4/5 interspace, below which anaesthetists avoids the termination of the spinal cord. The same blind "anatomical rule" is used throughout anaesthetics, whether the patient is male or female, young or old, pregnant or non-pregnant, supine or lateral, an approach that is clearly far from robust. The physiological changes of pregnancy such as fluid retention and weight gain can further make identification of the standard landmarks challenging. Advances in ultrasound technology have allowed direct visualisation of the bones in the back. Studies have shown that the conventional anatomical based method for locating the point of needle insertion is unreliable even amongst experienced anaesthetists.

Spinal or epidural anaesthesia can be performed with the patient either sitting or lying on their side. The investigators aim to determine whether a difference exists between the perceived mid-point of the L4/L5 intervertebral space, identified using manual demarcation of Tuffier's line, in these two positions. Ultrasound will then be used to ascertain the distance from the "true" midpoint.

ELIGIBILITY:
Inclusion Criteria:

* >37 weeks gestation
* BMI<40
* Singleton pregnancy
* Aged 16 to 65 years old.
* Latent phase of labour (<4cm cervix dilatation).

Exclusion Criteria:

* Previous spinal surgery
* Scoliosis
* Age<16
* Patient unable to tolerate positions
* Degenerative disease of the spine
* Patient refusal or inability to provide informed consent
* Patient in established labour (i.e. >4cm cervical dilatation)

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant parturients in the third trimester.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Discrepancy in distance between palpation vs. ultrasound midpoint of L4/5. interspace. | 15-30 minutes
  Distance (mm) between the mid-point of the L4/L5 intervertebral space in sitting and lateral decubitus positions, identified through manual palpation compared to the "true" mid-point measured by ultrasound.

SECONDARY OUTCOMES:
Discrepancy in distance between ultrasound midpoint of L4/5 in sitting vs. lateral position | 15-30 minutes
  Distance (mm) between the mid-point of the L4/L5 intervertebral space identified by ultrasound in sitting versus lateral decubitus positions.

CONTACTS AND LOCATIONS:
Overall Officials: Nhathien Nguyen-Lu, FRCA, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No